CLINICAL TRIAL: NCT05631236
Title: Promoting Cognitive Resilience and Reducing Frailty in Older Veterans With Bright Light Therapy
Acronym: Brite-VET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E4420-P; I21RX004420-01 (NIH)
Record Dates: First submitted 2022-08-09; First posted 2022-11-30 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Veteran Aged 65 and Older
Keywords: sleep; aging; veteran; cognition; dementia; functional capacity; frailty
MeSH Terms: conditions — Dementia; Frailty | interventions — Ultraviolet Therapy

STUDY DESIGN:
Intervention Model Description: Randomized placebo control trial.
Who Masked: Participant
Masking Description: Bright light therapy devices include two sets: intervention that emit blue light and the control that emits light at a non-therapeutic intensity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- BLT control (Placebo Comparator): Bright light glasses that emit a non-therapeutic blue light.
  Interventions: Device: Bright Light Therapy (AYO Glasses)
- BLT intervention (Active Comparator): Bright light glasses that emit a more intense therapeutic blue light.
  Interventions: Device: Bright Light Therapy (AYO Glasses)

INTERVENTIONS:
Device: Bright Light Therapy (AYO Glasses) — Bright light glasses that emit a more intense therapeutic blue light.
  Arms: BLT intervention
Device: Bright Light Therapy (AYO Glasses) — Bright light glasses that emit a non-therapeutic blue light.
  Arms: BLT control

SUMMARY:
Frailty is a multifactorial syndrome characterized by vulnerability to stressors that is intricately linked to cognitive impairment and mortality risk. Bright light therapy (BLT) reduces circadian disturbances by resynchronizing the hypothalamic biological clock via specific wavelengths of light. Human trials have demonstrated that BLT improves sleep quality and cognitive function in older adults. However, BLT has not been examined for use in older Veteran populations, particularly the impact on frailty. This randomized trial will assess the feasibility of employing BLT to study impacts on frailty, cognition, and sleep in older Veterans. Findings from this pilot will establish the power and effect size necessary for larger trials to support the use of BLT as readily available home-based treatment to improve healthspan of Veterans.

DETAILED DESCRIPTION:
Promoting cognition and reducing frailty in older Veterans with bright light therapy Frailty is a multifactorial syndrome characterized by vulnerability to stressors that increases disability and mortality risk. Thirty percent of Veterans 65 years or older are frail, which is three-times higher than aged matched non-Veterans. Frailty is intricately linked with cognitive impairment and Veterans are particularly susceptible with 14 percent exhibiting cognitive decline, some with early onset as young as 45 years of age. Importantly, 70% of frail and cognitively impaired older adults exhibit sleep disturbances, which makes identifying and improving sleep quality an attractive therapeutic strategy to enhance healthspan. Furthermore, this is of special interest as 55% of older Veterans experience sleep disturbances. The goal of this study is to examine the feasibility of utilizing bright light therapy (BLT) as a strategy to improve sleep via reduction of circadian rhythm disturbances. The long-term goal is to assess the potential for improving cognition and reducing frailty in older Veterans. BLT works by resynchronizing the hypothalamic biological clock via brief exposure to specific wavelengths of light following awakening, which restores melatonin and circadian rhythms. However, BLT has not been examined for reducing frailty in older Veteran populations. This project will therefore lay the foundation for larger trials the evaluate BLT in the treatment and prevention of cognitive disorders and to promote healthy aging.

ELIGIBILITY:
Inclusion Criteria:

* Participants studied in this project will include 30 men and 5 women of any race who are community dwellers
* The investigators seek to recruit relatively healthy individuals that may or may not exhibit early-stage co-morbidities

Exclusion Criteria:

* The investigators will exclude individuals without sleep disturbances (PSQI >5)
* Are morbidly obese (BMI > 40)
* Exhibit severe or advanced co-morbidities, or have cognitive impairment

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 30 men and 5 women
Enrollment: 43 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sleep quality | Change from baseline to endpoint at 12 weeks
  Sleep quality as assessed by Pittsburgh Sleep Quality Index (PSQI). The PSQI contains 19 self-rated questions that combined to form 7 component scores, each with a range of 0 to 3 points. These in turn are added to yield a global score with a range of 0 to 21 points. Higher scores indicate worse sleep quality.

SECONDARY OUTCOMES:
Short Physical Performance Battery | Change from baseline to endpoint at 12 weeks
  The Short physical performance battery (SPPB) is a battery of test often used in geriatric research to capture functional capacity in older adults. The test includes a balance and coordination assessment via asking participants to hold stances with three different foot positions (side-by-side, semi-tandem, and tandem: score 0-4), a gait speed test of approximately 10 feet (score 0-4 based on time), and a chair rise timed test where a participant is asked to rise from a chair 5 times (score 0-4 based on time). The composite score is therefore 0 to 12. Higher scores indicate better performance.
Frailty assessment | Change from baseline to endpoint at 12 weeks
  Frailty is a syndrome marked by greater susceptibility to adverse outcomes like falls and disability. We will be using the Fried Frailty Phenotype that includes: 1) unexpected weight loss of 5% or more in the last year or BMI < 18.5; score 0 or 1 if positive, 2) grip strength with BMI dependent cut points for men and women; score 0 or 1 if positive, 3) gait speed with height and sex dependent cutoffs; score 0 or 1 if positive, 4) activity assessed by a survey of the frequency of mild/moderate/energetic physical activity; score of 0 or 1, the latter if positive for hardly ever or never engaging in moderate or energetic physical activity, and 5) endurance assessed by survey of bed rest during the day; score of 0 or 1, the latter if occurring every day or every week. The composite score is therefore 0 to 5. Higher scores indicate more frailty.
Gait speed | Change from baseline to endpoint at 12 weeks
  Participants are asked to perform a timed walk of approximately 15 feet in length.
Muscle strength | Change from baseline to endpoint at 12 weeks
  Change from baseline to endpoint at 12 weeks Leg and arm strength will be measured using a small handheld dynamometer where the device is placed on the wrist or ankle as the participant is asked to extend or contract the limb with full force.
Body Composition (Lean and fat mass) | Change from baseline to endpoint at 12 weeks
  Body composition will be measured using bioelectric impedance (BIA) - a technique where participants are asked to stand on the measurement device and hold on to two metal handles. A light - and non-detectable - current is then transmitted allowing for collection of body fat and lean mass in the subject. The assessment takes roughly 2-3 minutes.
Interleukin-6 | Change from baseline at 12 weeks
  Chronic inflammation may be indicative of distress and lead to chronic diseases. The study will examine the change in interleukin-6 in picograms per milliliter in serum from baseline to endpoint at 12 weeks.
Sleep quantity | Change from baseline at 12 weeks
  Objectively measure sleep quantity using FITBIT Charge 5 devices. These devices are worn on the wrist and can measure total sleep time.
Step counts | Change from baseline to endpoint at 12 weeks
  Objectively measure activity using FITBIT Charge 5 actigraphy devices. These devices are worn on the wrist and capture total steps.
Cognitive screen - SLUMS | Change from baseline to endpoint at 12 weeks
  Cognitive status will be assessed using the VA - St. Louis University Mental Survey (VA-SLUMS) involving memory tests, shape recognition, and story recall. The survey scores range from 0 to 30, with a higher score representing greater cognitive capability.
Brain Derived Neurotrophic Factor (BDNF) | Change from baseline to endpoint at 12 weeks
  Serum cognitive marker: change in Brain Derived Neurotrophic Factor (BDNF) in picograms per milliliter from baseline to endpoint after 12 weeks.
Sleepiness | Change from baseline at 12 weeks
  Sleepiness as assessed by the Epworth Sleepiness Scale, which contains 8 self-rated questions with an aggregate score range of 0 to 24.
Fatigue | Change from baseline at 12 weeks
  Fatigue as assessed by the Brief Fatigue Inventory, which contains 9 self-rated questions with an aggregate score range of 0 to 90.
Sleep disorders | Change from baseline at 12 weeks
  Sleep disorders as assessed by the Holland Sleep Disorders Questionnaire, which contains 32 self-rated questions with an aggregate score range of 32 and 160. Higher scores indicate more sleep disorders.
Amyloid beta 42/40 ratio | Change from baseline at 12 weeks
  Serum cognitive marker: change in amyloid beta 42/40 ratio (a unitless measure derived from the ratio of serum amyloid-beta 42 in picograms per milliliter divided by serum amyloid-beta 40 in picograms per milliliter) from baseline to endpoint after 12 weeks.
Cognitive screen - Cognivue | Change from baseline at 12 weeks
  Cognivue to assess cognition. This is a computer based combinatorial visual and reaction time test, which is scored 0 to 100. Higher scores indicate better cognitive performance.
Sleep stages | Change from baseline to endpoint at 12 weeks
  Objectively measure duration of sleep stages using FITBIT Charge 5 devices. These devices are worn on the wrist and assess time spent in light, deep, and REM sleep stages.
Phosphorylated tau (P-tau) | Change from baseline at 12 weeks
  Serum cognitive marker: plasma levels of phosphorylated tau (P-tau) in picograms per milliliter from baseline to endpoint after 12 weeks.
Interleukin-10 | Change from baseline at 12 weeks
  Chronic inflammation may be indicative of distress and lead to chronic diseases. The study will examine the change in interleukin-10 in picograms per milliliter in serum from baseline to endpoint at 12 weeks.
Insomnia | Change from baseline at 12 weeks
  Insomnia as assessed by the Insomnia Severity Index, which contains 7 self-rated questions with an aggregate score range of 0 to 28.
Sleep chronotype | Change from baseline at 12 weeks
  Sleep chronotype as assessed by the Morningness/Eveningness survey, which contains 19 self-rated questions with an aggregate score range of 19 to 72.
Quality of life assessment | Change from baseline to endpoint at 12 weeks
  Change from baseline to endpoint at 12 weeks Quality of life assessment is performed using the Quality of life, enjoyment, and satisfaction questionnaire - short form (Q-LES-Q-SF) survey instrument. The survey instrument scores from 0 to 70 with a greater score representing better quality of life.
Anxiety and depression | Change from baseline at 12 weeks
  Anxiety and depression as assessed by the Hospital Anxiety and Depression Scale (HADS), which contains 14 self-rated questions with an aggregate score range of 0 to 21. Higher scores indicate greater anxiety and depression.
C-Reactive Protein | Change from baseline to endpoint at 12 weeks
  Chronic inflammation may be indicative of distress and lead to chronic diseases. The study will examine the change in C-reactive protein in picograms per milliliter in serum from baseline to endpoint at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce R. Troen, MD, Principal Investigator — Kansas City VA Medical Center, Kansas City, MO
Locations (1):
- Kansas City VA Medical Center, Kansas City, MO, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Final data sets will be made available upon specific request and under an authorized Data Use Agreement. This, in addition to the publications being made available via PubMed Central, will enable validation of results by recipients.
Supporting Information: Study Protocol
Time Frame: After analysis and completion of study along with subsequent publication of results.
Access Criteria: After analysis and completion of study along with subsequent publication of results.

DOCUMENTS (1):
  • Informed Consent Form (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT05631236/ICF_000.pdf